CLINICAL TRIAL: NCT03105115
Title: Effect of Intrathecal Fentanyl on Spinal Anesthesia During Dexmedetomidine
Brief Title: Effect of Intrathecal Fentanyl on Spinal Anesthesia During Dexmedetomidine Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1612-099-815
Record Dates: First submitted 2017-03-30; First posted 2017-04-07 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia, Spinal
Keywords: fentanyl; dexmedetomidine
MeSH Terms: interventions — Fentanyl; ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intrathecal fentanyl (Active Comparator): heavy bupivacaine 14mg and fentanyl 20mcg will be injected intrathecally during spinal anesthesia
  Interventions: Drug: fentanyl
- bupivacaine only (Experimental): heavy bupivacaine 14mg will be injected intrathecally during spinal anesthesia
  Interventions: Drug: bupivacaine only

INTERVENTIONS:
Drug: fentanyl — intrathecal fentanyl will be added as adjuvant for spinal anesthesia using heavy bupivacaine, while dexmedetomidine will be infused intravenously during operation
  Other Names: Hana Pharmacy
  Arms: intrathecal fentanyl
Drug: bupivacaine only — heavy bupivacaine will be injected intrathecally during spinal anesthesia, without fentanyl, while dexmedetomidine will be infused intravenously during operation
  Other Names: AstraZeneca
  Arms: bupivacaine only

SUMMARY:
Intravenous infusion of dexmedetomidine during procedure was known to be associated prolonged duration of spinal anesthesia. In patients receiving dexmedetomidine infusion during procedure, it has been not evaluated whether use of adjuvant intrathecal fentanyl had additional prolonging effect on duration of spinal anesthesia or not. Therefore, the investigators planned this trial to compare clinical outcomes in patients receiving spinal anesthesia with heavy bupivacaine only and heavy bupivacaine plus fentanyl adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing total knee replacement arthroplasty under spinal anesthesia

Exclusion Criteria:

* Contraindication of spinal anesthesia
* inability to communicate
* morbid obesity (BMI > 30kg/m2)
* spine abnormality
* severe cardiac dysfunction
* Height <155cm, or > 180cm
* contraindication to fentanyl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Two segment sensory block regression time | From completion of spinal anesthesia, to end of surgery, an expected average of 2 hours
  Time from highest sensory block level to two segment regression

SECONDARY OUTCOMES:
motor block | From completion of spinal anesthesia, to end of surgery, an expected average of 2 hours
  modified Bromage scale
postoperative pain score | at op day, at postoperative 1st day, at postoperative 2nd day
  VAS scale
postoperative nausea and vomiting | at op day, at postoperative 1st day, at postoperative 2nd day
  VAS scale
intraoperative incidence of hypotension | From completion of spinal anesthesia, to end of surgery, an expected average of 2 hours
  hypotension : SBP decreased by more than 30% of baseline SBP

CONTACTS AND LOCATIONS:
Overall Officials: Jin-tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seetharam KR, Bhat G. Effects of isobaric ropivacaine with or without fentanyl in subarachnoid blockade: A prospective double-blind, randomized study. Anesth Essays Res. 2015 May-Aug;9(2):173-7. doi: 10.4103/0259-1162.152149. PMID 26417123
- [Background] Singh R, Kundra S, Gupta S, Grewal A, Tewari A. Effect of clonidine and/or fentanyl in combination with intrathecal bupivacaine for lower limb surgery. J Anaesthesiol Clin Pharmacol. 2015 Oct-Dec;31(4):485-90. doi: 10.4103/0970-9185.169069. PMID 26702205
- [Derived] Park SK, Lee JH, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Comparison of bupivacaine plus intrathecal fentanyl and bupivacaine alone for spinal anesthesia with intravenous dexmedetomidine sedation: a randomized, double-blind, noninferiority trial. Reg Anesth Pain Med. 2019 Apr;44(4):459-465. doi: 10.1136/rapm-2018-100084. Epub 2019 Jan 23. PMID 30679336